CLINICAL TRIAL: NCT03090178
Title: Sleep & Quality of Life Evaluation of Patients With Atopic Dermatitis Based on Real-world Data Collection With a Smartphone Application and a Validated Actigraphy Wristband
Brief Title: Sleep & Quality of Life Evaluation of Patients With Atopic Dermatitis Based on E-diary on a Smartphone Application and Actigraphy
Acronym: ACTISLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: P004
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Intervention Model Description: Investigators will first enroll patients, then healthy volunters. Healthy volunters will be matched to patients on age, sexe and wake up at a programmed time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Wear a wristband actigraph while sleeping and answer to quality of questionnaires on a smartphone application:
  * sleep diary
  * Pruritus
  * dermatology life quality index
  Interventions: Other: electronic-Patient Report Outcome and wear of a wristband actigraph
- Healthy Volunteers (Active Comparator): Wear of a wristband actigraph while sleeping and answer to quality of questionnaires on a smartphone application:
  * sleep diary
  * Pruritus
  * dermatology life quality index
  Interventions: Other: electronic-Patient Report Outcome and wear of a wristband actigraph

INTERVENTIONS:
Other: electronic-Patient Report Outcome and wear of a wristband actigraph — Measurement of sleep quality and quantity with wristband actigraph and evaluation of quality of life with electronic-Patient Report Outcome

SUMMARY:
Atopic dermatitis is a chronic disease with a high impact on patient's quality of life. Nocturnal pruritus is one of the main symptoms affecting quality of life. Treatment efficacy is generally measured by healthcare professionals during consultations with both questioning and visual examination of the lesions. Quality of Life (QoL) can also be evaluated retrospectively with the Dermatology Life Quality Index (DLQI) scale. Collecting data retrospectively introduces a significant recall bias that can be addressed by collecting data in Real World (RW). Real World data collection is prospective and take place within the patient's own environment. While data collection is generally done with diaries, it has been demonstrated that smartphone and connected devices were able to produce more precise and granular data than traditional methods.

DETAILED DESCRIPTION:
The main objective of the study is to demonstrate a medical hypothesis using a wristband actigraph: patients with moderate to severe atopic dermatitis have a poorer quality and quantity of sleep than healthy subject.

Secondary objetives are to assess the interest of a smartphone application in evaluating the quality of life of patients with moderate to severe atopic dermatitis in regard of those of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Subjects using a smartphone running Apple operating system (iOS 7 and above) or Android (version 2.2 and above)
* Subjects agreeing to wear the actigraphy wristband at night
* Subjects 18 years old or older
* Subjects affiliated to French Health Insurance
* Subjects treated for moderate to severe atopic dermatitis or atopic dermatitis exacerbation* *The stage of the atopic dermatitis will be assessed by using the Eczema Area and Severity Index (EASI), Body Surface Area (BSA) and Investigator Global Assessment (IGA). The EASI is an investigator-assessed instrument measuring the severity of clinical signs in atopic dermatitis. The EASI was identified as one of the best-validated outcome measures for atopic dermatitis.

A moderate to severe atopic dermatitis corresponds to:

* Eczema Area and Severity Index score ≥ 7.1
* Investigator Global Assessment ≥ 3
* Body Surface Area ≥ 10

Healthy volunters :

* Subjects using a smartphone running iOS (iOS 7 and above) or Android (version 2.2 and above)
* Subjects agreeing to wear the actigraphy wristband at night
* Subjects 18 years old or older
* Subjects affiliated to French Health Insurance
* Subjects without a dermatology disease

Non inclusion Criteria:

* -Illiterate subjects
* Subjects not proficient in French
* Subject with a primary insomnia*

  *Insomnia, sleep apnea and hypersomnia will be evaluated with respectively 3 tests:
* Insomnia Severity Index (ISI);
* Berlin Sleep Apnea Scale;
* Epworth Scale
* Subjects treated by hypnotic drugs
* Pregnant woman
* Subjects under guardianship

Exclusion criteria:

If a participant is taking hypnotic treatments during his study participation, he will be excluded from the clinical trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 15 days
  Measure of sleep quality

SECONDARY OUTCOMES:
Sleep quantity | 15 days
  Measure of sleep quantity

OTHER OUTCOMES:
Quality of life | two times a day for 15 days
  electronic patient report outcome on a secured mobile application

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Louis, Paris, France